CLINICAL TRIAL: NCT01729091
Title: Phase II Study of Umbilical Cord Blood-Derived Natural Killer Cells in Conjunction With Elotuzumab, Lenalidomide and High Dose Melphalan Followed by Autologous Stem Cell Transplant for Patients With Multiple Myeloma
Brief Title: Umbilical Cord Blood-Derived Natural Killer Cells, Elotuzumab, Lenalidomide, and High Dose Melphalan, Followed by Stem Cell Transplant in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0379; NCI-2014-01096 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RV-MM-PI-0691; NCI-2014-00541; 2011-0379 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2012-11-09; First posted 2012-11-20 (Estimated); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Plasma Cell Leukemia; Plasma Cell Myeloma
MeSH Terms: conditions — Leukemia, Plasma Cell; Multiple Myeloma | interventions — elotuzumab; Lenalidomide; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemotherapy, UCB-derived NK cells, transplant) (Experimental): Patients receive elotuzumab IV over 2-5 hours on day -15 and -8, lenalidomide PO QD on days -8 to -2, high-dose melphalan IV over 30 minutes on day -7, and UCB-derived NK cells IV over 1 hour on day -5. Patients undergo autologous stem cell transplant on day 0.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Biological: Elotuzumab; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Drug: Melphalan; Biological: Natural Killer Cell Therapy; Biological: Umbilical Cord Blood-Derived Lymphocyte Therapy

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autologous stem cell transplant
  Other Names: Autologous Hematopoietic Cell Transplantation; autologous stem cell transplantation
Biological: Elotuzumab — Given IV
  Other Names: BMS-901608; Empliciti; HuLuc-63; HuLuc63; PDL-063; PDL063
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine nitrogen mustard; Sarcoclorin; Sarkolysin; WR-19813
Biological: Natural Killer Cell Therapy — Given IV
Biological: Umbilical Cord Blood-Derived Lymphocyte Therapy — Given IV

SUMMARY:
This phase II trial studies the side effects and best dose of umbilical cord blood-derived natural killer cells when given together with elotuzumab, lenalidomide, and high dose melphalan before autologous stem cell transplant and to see how well they work in treating patients with multiple myeloma. Before transplant, stem cells are taken from patients and stored. Immunotherapy with monoclonal antibodies, such as elotuzumab, may induce changes in the body's immune system and may interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as lenalidomide and melphalan, may work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy before a stem cell transplant stops the growth of cancer cells by stopping them from dividing or killing them. Giving natural killer cells from donor umbilical cord blood before transplant may also kill myeloma cells that remain in the body after the last chemotherapy treatment. After treatment, stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To find the maximum tolerated dose (MTD) of umbilical cord blood (UCB)-derived natural killer (NK) cells.

II. To determine efficacy by the percent of patients achieving very good partial remission (VGPR) + complete remission (CR) at 3 months post-transplant.

III. To assess the minimal residual disease rate 100 days post-transplant in high-risk patients.

SECONDARY OBJECTIVE:

I. To quantify duration of infused allogeneic donor UCB-derived NK cells in the recipient.

OUTLINE: This is a dose-escalation study of UCB-derived NK cells.

Patients receive elotuzumab intravenously (IV) over 2-5 hours on day -15 and -8, lenalidomide orally (PO) once daily (QD) on days -8 to -2, high-dose melphalan IV over 30 minutes on day -7, and UCB-derived NK cells IV over 1 hour on day -5. Patients undergo autologous stem cell transplant on day 0.

After completion of study treatment, patients are followed up at 30, 60 and 100 days and 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high risk multiple myeloma who are transplant candidates, in partial response (PR) or better; high risk will be defined as patients with any of the following:

  * Fluorescence in situ hybridization showing t(4:14), t(14:16), t(14:20), gain (amp) 1q; deletion (Del) 17/17p [or tp53 gene mutation/deletion by next generation sequencing (NGS), or by conventional cytogenetics];
  * Deletion 13 by conventional cytogenetic analysis;
  * High risk signatures as determined by the GEP-70 or EMC-92 gene expression profiles;
  * Relapsed disease within 18 months of prior autologous stem cell transplant (ASCT)
* Patients with plasma cell leukemia who are transplant candidates
* Performance score of at least 70% by Karnofsky or 0 to 2 Eastern Cooperative Oncology Group (ECOG)
* Left ventricular ejection fraction greater than 40%
* Pulmonary function test (PFT) demonstrating a diffusion capacity of least 40% predicted
* Estimated serum creatinine clearance >= 60 ml/min (using the Cockcroft-Gault formula and/or serum creatinine =< 1.6 mg/dL
* Serum glutamate pyruvate transaminase (SGPT) less than 3 x upper limit of normal
* Total bilirubin less than 2 x upper limit of normal
* All study participants must be registered into the mandatory Revlimid Risk Evaluation and Mitigation Strategy (REMS) program, and be willing and able to comply with the requirements of the Revlimid REMS program
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS program
* Men must agree to use a latex condom during sexual contact with females of child bearing potential even if they have had a successful vasectomy
* Patients must have a cord blood (CB) unit available which is matched with the patient at 4, 5, or 6/6 human leukocyte antigen (HLA) class I (serological) and II (molecular) antigens
* Patient or legally authorized representative able to sign informed consent

Exclusion Criteria:

* Patients receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to melphalan
* Known hypersensitivity or desquamating rash to either thalidomide or lenalidomide
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, uncontrolled hypertension (systolic > 160, diastolic > 100 despite antihypertensive therapy, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Human immunodeficiency virus (HIV)-positive patients are excluded due to increased risk of lethal infections when treated with myeloablative chemotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-06-10 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samer S Srour, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were registered in MD Anderson Cancer Center.
Groups:
- P1_C1_5x10^6; P1_C2_1x10^7; P1_C3_5x10^7; P1_C4_1X10^8: Patients receive lenalidomide PO QD on days -8 to -2, high-dose melphalan IV over 30 minutes on day -7, and UCB-derived NK cells IV over 1 hour on day -5. Patients undergo autologous stem cell transplant on day 0.
  Autologous Hematopoietic Stem Cell Transplantation: Undergo autologous stem cell transplant
  Elotuzumab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Lenalidomide: Given PO
  Melphalan: Given IV
  Natural Killer Cell Therapy: Given IV
  Umbilical Cord Blood-Derived Lymphocyte Therapy: Given IV
- P2_1x10^8+Elotuzumab: Patients receive elotuzumab IV over 2-5 hours on day -15 and -8, lenalidomide PO QD on days -8 to -2, high-dose melphalan IV over 30 minutes on day -7, and UCB-derived NK cells IV over 1 hour on day -5. Patients undergo autologous stem cell transplant on day 0.
  Autologous Hematopoietic Stem Cell Transplantation: Undergo autologous stem cell transplant
  Elotuzumab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Lenalidomide: Given PO
  Melphalan: Given IV
  Natural Killer Cell Therapy: Given IV
  Umbilical Cord Blood-Derived Lymphocyte Therapy: Given IV
Period: Overall Study
Arm/Group | P1_C1_5x10^6 | P1_C2_1x10^7 | P1_C3_5x10^7 | P1_C4_1X10^8 | P2_1x10^8+Elotuzumab
Started | 3 | 3 | 4 | 32 | 30
Completed | 3 | 3 | 4 | 32 | 30
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | P1_C1_5x10^6 | P1_C2_1x10^7 | P1_C3_5x10^7 | P1_C4_1X10^8 | P2_1x10^8+Elotuzumab | Total
Number analyzed (Participants) | 3 | 3 | 4 | 32 | 30 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3 | 26 | 21 | 53
  >=65 years | 1 | 2 | 1 | 6 | 9 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 14 | 7 | 24
  Male | 3 | 1 | 3 | 18 | 23 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 5 | 3 | 8
  Not Hispanic or Latino | 3 | 3 | 4 | 27 | 27 | 64
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 4 | 32 | 30 | 72

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: Dose limiting toxicity is defined as number of participants experienced:
  * grade 4 NK infusion related toxicity,
  * failure to engraft by D+28 or delayed engraftment,
  * grades 3-5 allergic reactions related to study cell infusion,
  * grade 3-5 organ toxicity (cardiac, dermatologic, gastrointestinal, hepatic, pulmonary, renal/genitourinary, or neurologic) not pre-existing or due to the underlying malignancy or due to preparative chemotherapy and occurring within 30 days (+3 days if necessary) post-transplant,
  * grades 3-4 acute GVHD occurring within 45 days post-transplant,
  * treatment-related death within 8 weeks of the study cell infusion.
Time Frame: Within 30 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | P1_C1_5x10^6 | P1_C2_1x10^7 | P1_C3_5x10^7 | P1_C4_1X10^8 | P2_1x10^8+Elotuzumab
Number analyzed (Participants) | 3 | 3 | 4 | 32 | 30
Participants
  grade 4 NK infusion related toxicity | 0 | 0 | 0 | 0 | 0
  failure to engraft by D+28 or delayed engraftment | 0 | 0 | 0 | 1 | 0
  · grades 3-5 allergic reactions related to study cell infusion | 0 | 0 | 0 | 0 | 0
  grade 3-5 organ toxicity | 1 | 0 | 0 | 13 | 11
  grades 3-4 acute GVHD occurring within 45 days post-transplant | 0 | 0 | 0 | 0 | 0
  treatment-related death within 8 weeks of the study cell infusion | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants That Achieved Very Good Response (VGPR) + Complete Response (CR)
Description: Complete response (CR) (all of the following):
  1. Negative immunofixation in serum and urine.
  2. < 5% plasma cells in the bone marrow.
  3. Disappearance of any soft tissue plasmacytomas.
  Very good partial response (VGPR) (one of the following):
  1. Serum and urine M protein detectable by immunofixation but not by electrophoresis.
  2. 90% or greater reduction in serum M protein plus urine M protein level <100 mg per 4h.
Time Frame: At 3 months post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | P1_C1_5x10^6 | P1_C2_1x10^7 | P1_C3_5x10^7 | P1_C4_1X10^8 | P2_1x10^8+Elotuzumab
Number analyzed (Participants) | 3 | 3 | 4 | 32 | 30
Participants
  VGPR | 1 | 0 | 1 | 4 | 5
  CR | 1 | 3 | 2 | 17 | 22

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Number of participants that are alive and disease free one year post transplant
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | P1_C1_5x10^6 | P1_C2_1x10^7 | P1_C3_5x10^7 | P1_C4_1X10^8 | P2_1x10^8+Elotuzumab
Number analyzed (Participants) | 3 | 3 | 4 | 32 | 30
Participants | 2 | 2 | 4 | 28 | 28

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | P1_C1_5x10^6 | P1_C2_1x10^7 | P1_C3_5x10^7 | P1_C4_1X10^8 | P2_1x10^8+Elotuzumab
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/3 | 2/4 | 11/32 | 3/30
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/4 | 1/32 | 1/30
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 32/32 | 27/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P1_C1_5x10^6 (N=3) | P1_C2_1x10^7 (N=3) | P1_C3_5x10^7 (N=4) | P1_C4_1X10^8 (N=32) | P2_1x10^8+Elotuzumab (N=30)
Low platelet (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Primary graft failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P1_C1_5x10^6 (N=3) | P1_C2_1x10^7 (N=3) | P1_C3_5x10^7 (N=4) | P1_C4_1X10^8 (N=32) | P2_1x10^8+Elotuzumab (N=30)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ALK increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
ALT increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 6 (6)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AST increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
Bacterial (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 8 (8) | 7 (7)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 3 (3) | 27 (27) | 25 (25)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ejection fraction decreased (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Engraftment syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (2) | 14 (14) | 16 (16)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 8 (8)
Fluid overload (General disorders) | 0 (0) | 2 (2) | 1 (1) | 6 (6) | 14 (14)
Gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 4 (4) | 32 (32) | 27 (27)
Oral mucositis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 19 (19) | 14 (14)
Peripheral neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 6 (6) | 5 (5)
T bilirubin increased (Investigations) | 2 (2) | 2 (2) | 1 (1) | 5 (5) | 3 (3)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 5 (5) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT01729091/Prot_SAP_000.pdf